CLINICAL TRIAL: NCT00550069
Title: Late Preterm Infants:Clinical Course and Outcome From Birth Through Out the First Year of Life.
Brief Title: Observational Study of Infants Born at 34 to 37 Weeks of Gestation Until the Age of 1 Year
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Iris Morag, Sheba Medical Cener
Other Study IDs: SHEBA-07-4821-IM-CTIL
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Respiratory Distress; Hypoglycemia; Feeding Intolerance; Jaundice; Hypothermia; Developmental Delay
Keywords: late preterm infants; near term infants; outcome
MeSH Terms: conditions — Dyspnea; Hypoglycemia; Jaundice; Hypothermia; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Late preterm infants are at an increased risk for short and long term morbidity (during the 1st year of life, their neurodevelopmental status may also be delayed as compared to infants born at term). The term "near term infants" is probably a deceiving one.

DETAILED DESCRIPTION:
The study will include all near term infants born at 3 Israeli medical centers during a one year period.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 34wks- 37wks
* Singleton
* Without chromosomal abnormalities or malformations

Exclusion Criteria:

* No chromosomal abnormalities
* Malformations

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants born at a gestational age of 34-37 weeks in 3 medical centers in Israel
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-12; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
neurodevelopmental, health and growth status in late preterm infants vs. controls within the first year of life | one year

CONTACTS AND LOCATIONS:
Overall Officials: Iris Morag, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel